CLINICAL TRIAL: NCT03509467
Title: Using MC1R Genotype to Impact Melanoma Risk Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Ponce Health Sciences University (Other); University of South Florida (Other); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-17984; MCC-19461 (Other: H. Lee Moffitt Cancer and Research Center)
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Melanoma (Skin); Squamous Cell Carcinoma; Squamous Cell Cancer; Skin Cancer; Basal Cell Carcinoma; Basal Cell Cancer
Keywords: skin cancer prevention; educational materials; skin cancer risk; questionnaire; MC1R genotype
MeSH Terms: conditions — Melanoma; Carcinoma, Squamous Cell; Neoplasms, Squamous Cell; Skin Neoplasms; Carcinoma, Basal Cell; Neoplasms, Basal Cell | interventions — Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Group A (Experimental): Intervention Group A: Non-Hispanic White Population
  Post determination of MC1R Genotypes, participants randomized to the intervention group, will receive personalized information about ways that they can protect themselves and their child from developing melanoma.
  By the end of the study, all participants will have had the opportunity to receive information about their inherited risk.
  Interventions: Behavioral: Personalized Information; Other: DNA Extraction Determination of MC1R Genotypes
- Intervention Group B (Experimental): Intervention Group B: Hispanic Population
  Post determination of MC1R Genotypes, participants randomized to the intervention group, will receive personalized information about ways that they can protect themselves and their child from developing melanoma.
  By the end of the study, all participants will have had the opportunity to receive information about their inherited risk.
  Interventions: Behavioral: Personalized Information; Other: DNA Extraction Determination of MC1R Genotypes
- Control Group A (Placebo Comparator): Control Group A: Non-Hispanic White Population
  Post determination of MC1R Genotypes, participants randomized to the control group, you will receive standard information about ways that they can protect themselves and their child from developing melanoma.
  By the end of the study, all participants will have had the opportunity to receive information about their inherited risk. Participants randomized into the control group, by the end of the study will also have had the opportunity to receive personalized information about ways they can protect themselves and their child from developing melanoma.
  Interventions: Behavioral: Standard Information; Other: DNA Extraction Determination of MC1R Genotypes
- Control Group B (Placebo Comparator): Control Group B: Hispanic Population
  Post determination of MC1R Genotypes, participants randomized to the control group, you will receive standard information about ways that they can protect themselves and their child from developing melanoma.
  By the end of the study, all participants will have had the opportunity to receive information about their inherited risk. Participants randomized into the control group, by the end of the study will also have had the opportunity to receive personalized information about ways they can protect themselves and their child from developing melanoma.
  Interventions: Behavioral: Standard Information; Other: DNA Extraction Determination of MC1R Genotypes

INTERVENTIONS:
Behavioral: Personalized Information — Personalized information about ways that participants can protect themselves and their child from developing melanoma.
  Other Names: educational materials
  Arms: Intervention Group A; Intervention Group B
Behavioral: Standard Information — Standard information about ways that participants can protect themselves and their child from developing melanoma.
  Other Names: educational materials
  Arms: Control Group A; Control Group B
Other: DNA Extraction Determination of MC1R Genotypes — After signing informed consent, a biologic sample (saliva) will be collected for the purpose of DNA extraction determination of MC1R genotypes. All participants who carry high risk MC1R genotypes and a proportion of those who carry low risk or no MC1R variants will be randomized to the control or intervention arm.
  Other Names: risk factor

SUMMARY:
The purpose of this study is to examine how different messages about risk of melanoma can impact the way people protect themselves against developing these diseases.

ELIGIBILITY:
Inclusion Criteria:

CRITERIA FOR: NON-HISPANIC WHITE POPULATION

* Investigators will recruit participants from the Family Medicine and General Internal Medicine clinics of the Morsani Center at the University of South Florida.
* White, non-Hispanic patients who self-report a low phenotypic risk profile for development of melanoma and are able to read and speak English fluently.
* 18 years of age or older
* Capable of giving informed consent
* Potential participants will be screened for eligibility based on responses to questions about skin phenotypes, early detection behaviors and past history of melanoma.
* After signing informed consent, a biologic sample (saliva) will be collected for the purpose of DNA extraction determination of MC1R genotypes. All participants who carry high risk MC1R genotypes and a proportion of those who carry low risk or no MC1R variants will be randomized to the control or intervention arm.

CRITERIA FOR: HISPANIC POPULATION

* Investigators will recruit participants living in Tampa Bay and Puerto Rico as part of the U54 Ponce Health Sciences University-Moffitt Cancer Center (PHSU-MCC) Partnership. In Tampa Bay, participants will be recruited from the Family Medicine and General Internal Medicine clinics of the Morsani Center at the University of South Florida, and from the Suncoast Community Health Centers.
* Patients who self-report as Hispanics and are able to read and speak either Spanish or English fluently.
* 18 years of age or older
* Capable of giving informed consent
* Potential participants will be screened for eligibility based on responses to early detection behaviors and past history of melanoma.
* After signing informed consent, a biologic sample (saliva) will be collected for the purpose of DNA extraction determination of MC1R genotypes. All participants who carry high risk MC1R genotypes and a proportion of those who carry low risk or no MC1R variants will be randomized to the control or intervention arm.

Exclusion Criteria:

CRITERIA FOR: NON-HISPANIC WHITE POPULATION

* Have had a skin examination within the past year.
* Do not meet race/ethnicity criteria for their group
* White, non-Hispanic group - participants reporting sun-sensitive phenotypes
* A personal history of melanoma

CRITERIA FOR: HISPANIC POPULATION

* Have had a skin examination within the past year.
* Do not meet ethnicity criteria for their group
* White, non-Hispanic group - participants reporting sun-sensitive phenotypes
* Participants with a personal history of melanoma and/or more personal history of more than on squamous cell cancer (SCC) and/or Basal Cell Cancer (BCC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2054 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kanetsky, Ph.D, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States
- Ponce School of Medicine, Ponce, Puerto Rico

REFERENCES:
- [Derived] Rivera Rivera JN, Lacson JCA, Kim Y, Roetzheim RG, Sutton SK, Soto-Torres B, Vadaparampil ST, Kanetsky PA. Sharing and seeking information about skin cancer risk and prevention among Hispanic people from Florida and Puerto Rico. PEC Innov. 2023 Nov 14;3:100232. doi: 10.1016/j.pecinn.2023.100232. eCollection 2023 Dec 15. PMID 38028436
- [Derived] Lacson JCA, Sutton SK, Kim Y, Roetzheim RG, Vadaparampil ST, Soto-Torres B, Kanetsky PA. Predictors of correct recall of genetic risk information among Hispanic individuals in Florida and Puerto Rico. Patient Educ Couns. 2023 Dec;117:107978. doi: 10.1016/j.pec.2023.107978. Epub 2023 Sep 11. PMID 37708699
- [Derived] Lacson JCA, Kim Y, Roetzheim RG, Sutton SK, Vadaparampil ST, Kanetsky PA. Predictors of genetic risk recall among the participants of a randomized controlled precision prevention trial against melanoma. Genet Med. 2023 Apr;25(4):100005. doi: 10.1016/j.gim.2023.100005. Epub 2023 Jan 7. PMID 36629029
- [Derived] Lacson JCA, Doyle SH, Del Rio J, Forgas SM, Carvajal R, Gonzalez-Calderon G, Feliciano AR, Kim Y, Roetzheim RG, Sutton SK, Vadaparampil ST, Soto-Torres B, Kanetsky PA. A randomized clinical trial of precision prevention materials incorporating MC1R genetic risk to improve skin cancer prevention activities among Hispanics. Cancer Res Commun. 2022 Jan;2(1):28-38. doi: 10.1158/2767-9764.crc-21-0114. Epub 2022 Jan 11. PMID 35845857
- [Derived] Lacson JCA, Forgas SM, Doyle SH, Qian L, Del Rio J, Valavanis S, Carvajal R, Gonzalez-Calderon G, Kim Y, Roetzheim RG, Vadaparampil ST, Kanetsky PA. Assessment of melanoma precision prevention materials incorporating MC1R genetic risk information. Transl Behav Med. 2022 May 26;12(5):683-687. doi: 10.1093/tbm/ibac034. PMID 35552458

RESULTS

PARTICIPANT FLOW:
Groups:
- MC1R Average Risk- Control- Non-Hispanic White Population; MC1R Average Risk- Control- Hispanic Population: Post determination of MC1R Genotypes, participants in the average risk standard arm (control) received mailed materials containing information on (1) melanoma and skin cancer; and (2) melanoma prevention behaviors recommended by the American Academy of Dermatology. All participants received information on sun protection behaviors targeted at children.
- MC1R Average Risk - Intervention- Non-Hispanic White Population; MC1R Higher Risk - Intervention- Non-Hispanic White Population; MC1R Average Risk - Intervention- Hispanic Population; MC1R Higher Risk - Intervention- Hispanic Population: Post determination of MC1R Genotypes, participants in the average risk precision prevention arm (intervention) received mailed materials containing information on: (1) melanoma and skin cancer; (2) genetic risk for melanoma; (3) MC1R and its role in developing melanoma, their MC1R risk group, and interpretation of risk information; and (4) melanoma prevention behaviors in the context of genetic risk. All participants received information on sun protection behaviors targeted at children.
- MC1R Higher Risk- Control - Non-Hispanic White Population; MC1R Higher Risk- Control - Hispanic Population: Post determination of MC1R Genotypes, participants in the higher risk standard arm (control) received mailed materials containing information on (1) melanoma and skin cancer; and (2) melanoma prevention behaviors recommended by the American Academy of Dermatology. All participants received information on sun protection behaviors targeted at children.
Period: Overall Study
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Started | 227 | 226 | 339 | 342 | 195 | 195 | 262 | 268
Completed | 222 | 225 | 331 | 333 | 184 | 185 | 251 | 257
Not Completed | 5 | 1 | 8 | 9 | 11 | 10 | 11 | 11
Not completed — Withdrawal by Subject | 5 | 1 | 6 | 7 | 10 | 10 | 10 | 10
Not completed — Death | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 0
Not completed — Proxy Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants with at least one child ages 10 years of age or younger completed additional questions about the child's primary prevention activities
Groups:
- MC1R Average Risk - Intervention- Non-Hispanic White Population; MC1R Average Risk - Intervention- Hispanic Population: Participants in the average risk precision prevention arm (intervention) received mailed materials containing information on: (1) melanoma and skin cancer; (2) genetic risk for melanoma; (3) MC1R and its role in developing melanoma, their MC1R risk group, and interpretation of risk information; and (4) melanoma prevention behaviors in the context of genetic risk.
- MC1R Higher Risk - Intervention- Non-Hispanic White Population; MC1R Higher Risk - Intervention- Hispanic Population: Participants in the higher risk precision prevention arm (intervention) received mailed materials containing information on: (1) melanoma and skin cancer; (2) genetic risk for melanoma; (3) MC1R and its role in developing melanoma, their MC1R risk group, and interpretation of risk information; and (4) melanoma prevention behaviors in the context of genetic risk.
- Total: Total of all reporting groups
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population | Total
Number analyzed (Participants) | 227 | 226 | 339 | 342 | 195 | 195 | 262 | 268 | 2054
Age, Customized [Count of Participants; unit: Participants]
  Age <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 189 | 190 | 277 | 300 | 163 | 172 | 227 | 236 | 1754
  > =65 years | 38 | 36 | 62 | 42 | 32 | 22 | 35 | 31 | 298
  Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 115 | 110 | 164 | 174 | 55 | 58 | 66 | 79 | 821
  Female | 112 | 116 | 175 | 168 | 138 | 134 | 193 | 186 | 1222
  Unknown | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 195 | 195 | 262 | 268 | 920
  Not Hispanic or Latino | 227 | 226 | 339 | 342 | 0 | 0 | 0 | 0 | 1134
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 8
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 15 | 15 | 6 | 13 | 49
  White | 227 | 226 | 339 | 342 | 149 | 152 | 221 | 213 | 1869
  More than one race | 0 | 0 | 0 | 0 | 5 | 4 | 4 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 25 | 23 | 28 | 29 | 105
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 0 | 0 | 0 | 0 | 93 | 93 | 123 | 124 | 433
  United States | 227 | 226 | 339 | 342 | 102 | 102 | 139 | 144 | 1621

OUTCOME MEASURES:

1. Primary Outcome: Weekday Sun Exposure - NHW - Baseline
Description: Self-reported average hours spent outside during weekdays for the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
Hours | 1.27 (0.03) | 1.30 (0.03) | 1.26 (0.03) | 1.29 (0.03)

2. Primary Outcome: Weekday Sun Exposure - NHW - After Intervention
Description: Self-reported average hours spent outside during weekdays for the Non-Hispanic White Population after they received the intervention
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
Hours | 1.09 (0.04) | 1.18 (0.06) | 1.09 (0.05) | 1.05 (0.05)

3. Primary Outcome: Weekend Sun Exposure - NHW - Baseline
Description: Self-reported average hours spent outside during weekends for the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
Hours | 2.17 (0.04) | 2.25 (0.07) | 2.25 (0.04) | 2.30 (0.07)

4. Primary Outcome: Weekend Sun Exposure - NHW - After Intervention
Description: Self-reported average hours spent outside during weekends for the Non-Hispanic White Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
Hours | 2.00 (0.08) | 2.08 (0.07) | 1.89 (0.07) | 1.89 (0.07)

5. Primary Outcome: Sunburns - NHW - Baseline
Description: Self-reported number of red or painful sunburns for the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Sunburns
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
Sunburns | 0.60 (0.03) | 0.66 (0.04) | 0.83 (0.06) | 0.85 (0.06)

6. Primary Outcome: Sunburns - NHW - After Intervention
Description: Self-reported number of red or painful sunburns for the Non-Hispanic White Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Sunburns
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
Sunburns | 0.29 (0.04) | 0.20 (0.04) | 0.27 (0.04) | 0.28 (0.05)

7. Primary Outcome: Outdoor Intentional Tanning - NHW - Baseline
Description: Self-reported number on a scale from 1=never to 5=always for outdoor intentional tanning for the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
score on a scale | 2.01 (0.06) | 2.03 (0.06) | 1.96 (0.02) | 1.95 (0.02)

8. Primary Outcome: Outdoor Intentional Tanning - NHW - After Intervention
Description: Self-reported number on a scale from 1=never to 5=always outdoor intentional tanning for the Non-Hispanic White Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
score on a scale | 1.79 (0.07) | 1.82 (0.07) | 1.70 (0.04) | 1.71 (0.03)

9. Primary Outcome: Proportion of Participants Wearing a Hat - NHW - Baseline
Description: Proportion who practiced wearing a hat for the Non-Hispanic White Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: proportion of participants
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
proportion of participants | 0.20 (0.03) | 0.17 (0.03) | 0.25 (0.03) | 0.27 (0.03)

10. Primary Outcome: Proportion of Participants Wearing a Hat - NHW - After Intervention
Description: as for outcome 9
Time Frame: 12 Months
Measure: Mean (Standard Error); unit: proportion of participants
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
proportion of participants | 0.24 (0.04) | 0.29 (0.04) | 0.33 (0.03) | 0.32 (0.03)

11. Primary Outcome: Seeking Shade - NHW - Baseline
Description: Self-reported number of hours for seeking shade or using an umbrella outdoors for the Non-Hispanic White Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
Hours | 0.35 (0.04) | 0.27 (0.04) | 0.33 (0.03) | 0.34 (0.03)

12. Primary Outcome: Seeking Shade - NHW - After Intervention
Description: Self-reported number of hours for seeking shade or using an umbrella outdoors for the Non-Hispanic White Population after receiving the intervention. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: 12 Months
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
Hours | 0.34 (0.04) | 0.35 (0.04) | 0.35 (0.03) | 0.43 (0.03)

13. Primary Outcome: Wearing a Shirt - NHW - Baseline
Description: Self-reported number of hours for wearing a shirt with sleeves outdoors for the Non-Hispanic White Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
Hours | 0.72 (0.04) | 0.70 (0.04) | 0.68 (0.03) | 0.70 (0.03)

14. Primary Outcome: Wearing a Shirt - NHW - After Intervention
Description: Self-reported number of hours wearing a shirt with sleeves outdoors for the Non-Hispanic White Population after receiving the intervention. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: 12 Months
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
Hours | 0.71 (0.03) | 0.72 (0.03) | 0.67 (0.03) | 0.75 (0.02)

15. Primary Outcome: Wearing Sunglasses - NHW - Baseline
Description: Self-reported number of hours for wearing sunglasses outdoors for the Non-Hispanic White Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
Hours | 0.76 (0.03) | 0.75 (0.04) | 0.66 (0.03) | 0.70 (0.03)

16. Primary Outcome: Wearing Sunglasses - NHW - After Intervention
Description: Self-reported number of hours wearing sunglasses outdoors for the Non-Hispanic White Population after receiving the intervention. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: 12 Months
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
Hours | 0.77 (0.03) | 0.76 (0.04) | 0.70 (0.03) | 0.73 (0.03)

17. Primary Outcome: Wearing Sunscreen - NHW - Baseline
Description: Self-reported number of hours for wearing sunscreen outdoors for the Non-Hispanic White Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
Hours | 0.36 (0.04) | 0.28 (0.04) | 0.36 (0.04) | 0.40 (0.04)

18. Primary Outcome: Wearing Sunscreen - NHW - After Intervention
Description: Self-reported number of hours wearing sunscreen outdoors for the Non-Hispanic White Population after receiving the intervention. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: 12 Months
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
Hours | 0.36 (0.04) | 0.30 (0.04) | 0.42 (0.03) | 0.38 (0.03)

19. Primary Outcome: Participants With Indoor Intentional Tanning - NHW - Baseline
Description: Participants with at least one indoor intentional tanning session for the Non-Hispanic White Population
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 227 | 226 | 339 | 342
Participants | 10 | 12 | 18 | 7

20. Primary Outcome: Participants With Indoor Intentional Tanning - NHW - After Intervention
Description: Participants with at least one indoor intentional tanning session for the Non-Hispanic White Population after receiving the intervention
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 222 | 225 | 331 | 333
Participants | 4 | 9 | 15 | 7

21. Primary Outcome: Weekday Sun Exposure - Hispanic Population Baseline
Description: Self-reported number of hours of weekday sun exposure for the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
Hours | 1.70 (0.11) | 1.60 (0.11) | 1.74 (0.06) | 1.65 (0.05)

22. Primary Outcome: Weekday Sun Exposure - Hispanic Population After Intervention
Description: Self-reported number of hours of weekday sun exposure of the Hispanic population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
Hours | 1.38 (0.10) | 1.28 (0.10) | 1.38 (0.10) | 1.45 (0.10)

23. Primary Outcome: Weekend Sun Exposure - Hispanic Population - Baseline
Description: Self-reported number of hours of weekend sun exposure for the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
Hours | 2.04 (0.12) | 1.88 (0.11) | 2.05 (0.07) | 1.95 (0.07)

24. Primary Outcome: Weekend Sun Exposure - Hispanic Population - After Intervention
Description: Self-reported number of hours of weekend sun exposure for the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
Hours | 1.57 (0.10) | 1.62 (0.11) | 1.67 (0.07) | 1.57 (0.08)

25. Primary Outcome: Sunburns - Hispanic Population - Baseline
Description: Self-reported number of Sunburns for the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Sunburns
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
Sunburns | 0.42 (0.07) | 0.52 (0.07) | 0.47 (0.05) | 0.56 (0.05)

26. Primary Outcome: Sunburns - Hispanic Population - After Intervention
Description: Self-reported number of Sunburns for the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Sunburns
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
Sunburns | 0.10 (0.04) | 0.15 (0.05) | 0.21 (0.04) | 0.21 (0.04)

27. Primary Outcome: Outdoor Intentional Tanning - Hispanic Population - Baseline
Description: Self-reported number on a scale from 1=never to 5=always intentional tanning for the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
score on a scale | 1.64 (0.06) | 1.75 (0.07) | 1.64 (0.05) | 1.66 (0.05)

28. Primary Outcome: Outdoor Intentional Tanning - Hispanic Population - After Intervention
Description: Self-reported number on a scale from 1=never to 5=always outdoor intentional tanning for the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
score on a scale | 1.48 (0.05) | 1.49 (0.07) | 1.49 (0.05) | 1.48 (0.04)

29. Primary Outcome: Proportion of Participants Wearing a Hat - Hispanic Population - Baseline
Description: Proportion who practiced wearing a hat Often to Always for the Hispanic Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: proportion of participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
proportion of participants | 0.15 (0.03) | 0.12 (0.03) | 0.25 (0.04) | 0.17 (0.03)

30. Primary Outcome: Proportion of Participants Wearing a Hat - Hispanic Population - After Intervention
Description: Proportion who practiced wearing a hat Often to Always for the Hispanic Population after receiving the intervention. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: 9 months
Measure: Mean (Standard Error); unit: proportion of participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
proportion of participants | 0.19 (0.04) | 0.17 (0.03) | 0.32 (0.05) | 0.23 (0.04)

31. Primary Outcome: Seeking Shade - Hispanic Population - Baseline
Description: Self-reported number of hours of seeking shade or using an umbrella for the Hispanic Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
Hours | 0.42 (0.04) | 0.35 (0.03) | 0.43 (0.04) | 0.38 (0.03)

32. Primary Outcome: Seeking Shade - Hispanic Population - After Intervention
Description: Self-reported number of hours of seeking shade or using an umbrella for the Hispanic Population after receiving the intervention. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: 9 Months
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
Hours | 0.52 (0.04) | 0.46 (0.04) | 0.50 (0.06) | 0.53 (0.06)

33. Primary Outcome: Wearing a Shirt - Hispanic Population - Baseline
Description: Self-reported number of hours of wearing a shirt for the Hispanic Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
Hours | 0.66 (0.04) | 0.65 (0.04) | 0.70 (0.04) | 0.67 (0.04)

34. Primary Outcome: Wearing a Shirt - Hispanic Population - After Intervention
Description: Self-reported number of hours of wearing a shirt with sleeves outdoors for the Hispanic Population after receiving the intervention. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: 9 Months
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
Hours | 0.65 (0.04) | 0.63 (0.04) | 0.68 (0.04) | 0.72 (0.04)

35. Primary Outcome: Wearing Sunglasses - Hispanic Population - Baseline
Description: Self-reported number of hours of wearing sunglasses for the Hispanic Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
Hours | 0.52 (0.04) | 0.46 (0.04) | 0.54 (0.05) | 0.51 (0.04)

36. Primary Outcome: Wearing Sunglasses - Hispanic Population - After Intervention
Description: Self-reported number of hours of wearing sunglasses for the Hispanic Population after receiving the intervention. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: 9 Months
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
Hours | 0.52 (0.04) | 0.49 (0.04) | 0.54 (0.12) | 0.66 (0.10)

37. Primary Outcome: Wearing Sunscreen - Hispanic Population - Baseline
Description: Self-reported number of hours of wearing sunscreen for the Hispanic Population. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
Hours | 0.24 (0.03) | 0.16 (0.03) | 0.13 (0.02) | 0.15 (0.02)

38. Primary Outcome: Wearing Sunscreen - Hispanic Population - After Intervention
Description: Self-reported number of hours of wearing sunscreen for the Hispanic Population after receiving the intervention. This is a population predicted marginal proportion estimated by running a generalized estimating equation with the outcome modeled as a repeated binomial distribution (practiced the behavior often to always vs. sometimes, rarely, or never measured at both follow-ups) and using a logit link function. The model covariates included the baseline measure, any imbalanced baseline measures, predictors of missingness, and predictors of outcome.
Time Frame: 9 Months
Measure: Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
Hours | 0.25 (0.04) | 0.19 (0.03) | 0.13 (0.04) | 0.24 (0.06)

39. Primary Outcome: Participants With Intentional Indoor Tanning - Hispanic Population - Baseline
Description: Participants with at least one indoor intentional tanning session for the Hispanic Population
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 195 | 195 | 262 | 268
Participants | 4 | 6 | 5 | 7

40. Primary Outcome: Participants With Intentional Indoor Tanning - Hispanic Population - After Intervention
Description: Participants with at least one indoor intentional tanning session for the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 184 | 185 | 251 | 257
Participants | 3 | 2 | 6 | 5

41. Secondary Outcome: Weekday Sun Exposure - NHW Children - Baseline
Description: Self-reported average hours spent outside during weekdays among the children of the participants in the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 1.31 (0.09) | 1.50 (0.10) | 1.42 (0.08) | 1.40 (0.06)

42. Secondary Outcome: Weekday Sun Exposure - NHW Children - After Intervention
Description: as for outcome 41
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 1.29 (0.10) | 1.23 (0.14) | 1.34 (0.10) | 1.47 (0.10)

43. Secondary Outcome: Weekend Sun Exposure - NHW Children - Baseline
Description: Self-reported average hours spent outside during weekends among the children of the participants in the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 2.23 (0.07) | 2.29 (0.09) | 2.33 (0.08) | 2.26 (0.06)

44. Secondary Outcome: Weekend Sun Exposure - NHW Children - After Intervention
Description: as for outcome 43
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 2.36 (0.17) | 2.10 (0.17) | 2.28 (0.14) | 2.24 (0.14)

45. Secondary Outcome: Sunburns - NHW Children - Baseline
Description: Self-reported number of red or painful sunburns among the children of the participants in the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Sunburns
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Sunburns | 0.31 (0.08) | 0.48 (0.13) | 0.32 (0.04) | 0.37 (0.06)

46. Secondary Outcome: Sunburns - NHW Children - After Intervention
Description: Self-reported number of red or painful sunburns among the children of the participants in the Non-Hispanic White Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Sunburns
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Sunburns | 0.25 (0.11) | 0.16 (0.09) | 0.26 (0.04) | 0.10 (0.05)

47. Secondary Outcome: Outdoor International Tanning - NHW Children - Baseline
Description: Self-reported number of hours for outdoor intentional tanning among the children of the participants in the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 1.09 (0.06) | 1.13 (0.09) | 1.16 (0.03) | 1.10 (0.03)

48. Secondary Outcome: Outdoor Intentional Tanning - NHW Children - After Intervention
Description: Self-reported number of hours for outdoor intentional tanning among the children of the participants in the Non-Hispanic White Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 1.06 (0.05) | 0.99 (0.05) | 1.03 (0.03) | 1.06 (0.01)

49. Secondary Outcome: Wearing a Hat - NHW Children - Baseline
Description: Self-reported number of hours for wearing a hat outdoors among the children of the participants in the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 0.24 (0.09) | 0.11 (0.05) | 0.07 (0.02) | 0.09 (0.03)

50. Secondary Outcome: Wearing a Hat - NHW Children - After Intervention
Description: Self-reported number of hours for wearing a hat outdoors among the children of the participants in the Non-Hispanic White Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 0.08 (0.08) | 0.02 (0.03) | 0.07 (0.05) | 0.05 (0.04)

51. Secondary Outcome: Seeking Shade - NHW Children - Baseline
Description: Self-reported number of hours for seeking shade or using an umbrella outdoors among the children of the participants in the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 0.12 (0.07) | 0.19 (0.17) | 0.14 (0.04) | 0.15 (0.05)

52. Secondary Outcome: Seeking Shade - NHW Children - After Intervention
Description: Self-reported number of hours for seeking shade or using an umbrella outdoors among the children of the participants in the Non-Hispanic White Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 0.49 (0.26) | 0.17 (0.11) | 0.07 (0.04) | 0.18 (0.06)

53. Secondary Outcome: Wearing a Shirt - Average Risk NHW Children - Baseline
Description: Average Risk Participants children who wore a shirt with sleeves outdoors among the participants in the Non-Hispanic White Population
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21
Participants | 22 | 16

54. Secondary Outcome: Wearing a Shirt - Average Risk NHW Children - After Intervention
Description: as for outcome 53
Time Frame: 12 Month
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21
Participants | 25 | 21

55. Secondary Outcome: Wearing a Shirt - High Risk NHW Children - Baseline
Description: Self-reported number of hours wearing a shirt with sleeves outdoors among the children of the participants in the Non-Hispanic White High Risk Population
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 49 | 46
Hours | 0.91 (0.03) | 0.84 (0.04)

56. Secondary Outcome: Wearing a Shirt - High Risk NHW Children - After Intervention
Description: Self-reported number of hours wearing a shirt with sleeves outdoors among the children of the participants in the Non-Hispanic White High Risk Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 49 | 46
Hours | 0.85 (0.06) | 0.96 (0.03)

57. Secondary Outcome: Wearing Sunglasses - Average Risk NHW Children - Baseline
Description: Self-reported number of hours for wearing sunglasses outdoors among the children of the participants in the Non-Hispanic White Average Risk Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21
Hours | 0.04 (0.03) | 0.04 (0.03)

58. Secondary Outcome: Wearing Sunglasses - Average Risk NHW Children - After Intervention
Description: Self-reported number of hours wearing sunglasses outdoors among the children of the participants in the Non-Hispanic White Average Risk Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21
Hours | 0.01 (0.02) | 0.04 (0.06)

59. Secondary Outcome: Wearing Sunglasses -High Risk NHW Children - Baseline
Description: Children of the participants in the Non-Hispanic White High Risk Population who wore sunglasses outdoors
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 49 | 46
Participants | 3 | 7

60. Secondary Outcome: Wearing Sunglasses - High Risk NHW Children - After Intervention
Description: Children of the participants in the Non-Hispanic White High Risk Population who wore sunglasses outdoors after receiving the intervention
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 49 | 46
Participants | 4 | 7

61. Secondary Outcome: Wearing Sunscreen - NHW Children - Baseline
Description: Self-reported number of hours for wearing sunscreen outdoors among the children of the participants in the Non-Hispanic White Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 0.71 (0.08) | 0.66 (0.11) | 0.83 (0.04) | 0.88 (0.04)

62. Secondary Outcome: Wearing Sunscreen - NHW Children - After Intervention
Description: Self-reported number of hours wearing sunscreen outdoors among the children of the participants in the Non-Hispanic White Population after receiving the intervention
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population
Number analyzed (Participants) | 25 | 21 | 49 | 46
Hours | 0.70 (0.12) | 0.44 (0.24) | 0.69 (0.11) | 0.86 (0.06)

63. Secondary Outcome: Weekday Sun Exposure - Hispanic Children Population Baseline
Description: Self-reported number of hours of weekday sun exposure among the children of the participants in the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 1.48 (0.01) | 1.49 (0.02) | 1.73 (0.23) | 1.53 (0.18)

64. Secondary Outcome: Weekday Sun Exposure - Hispanic Children Population After Intervention
Description: Self-reported number of hours of weekday sun exposure among the children of the participants in the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 1.33 (0.09) | 1.04 (0.28) | 2.46 (0.29) | 0.90 (0.22)

65. Secondary Outcome: Weekend Sun Exposure - Hispanic Children Population - Baseline
Description: Self-reported number of hours of weekend sun exposure among the children of the participants in the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 1.80 (0.15) | 2.18 (0.13) | 1.87 (0.08) | 1.88 (0.08)

66. Secondary Outcome: Weekend Sun Exposure - Hispanic Children Population - After Intervention
Description: Self-reported number of hours of weekend sun exposure among the children of the participants in the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 1.56 (0.07) | 1.48 (0.12) | 2.18 (0.30) | 0.84 (0.39)

67. Secondary Outcome: Sun Protection Behaviors - Hispanic Children Population - Baseline
Description: Self-reported number of hours of sun protection behaviors among the children of the participants in the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 1.44 (0.16) | 1.51 (0.14) | 1.50 (0.03) | 1.55 (0.02)

68. Secondary Outcome: Sun Protection Behaviors - Hispanic Children Population - After Intervention
Description: Self-reported number of hours of sun protection behaviors among the children of the participants in the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 1.21 (0.28) | 1.68 (0.23) | 1.13 (0.17) | 1.98 (0.31)

69. Secondary Outcome: Outdoor Intentional Tanning - Hispanic Children Population - Baseline
Description: Self-reported number of hours of outdoor intentional tanning among the children of the participants in the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 1.43 (0.09) | 1.39 (0.09) | 1.24 (0.03) | 1.22 (0.02)

70. Secondary Outcome: Outdoor Intentional Tanning - Hispanic Children Population - After Intervention
Description: Self-reported number of hours of outdoor intentional tanning among the children of the participants in the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 0.93 (.39) | 1.64 (0.11) | 1.35 (0.15) | 1.06 (0.12)

71. Secondary Outcome: Sunburns - Hispanic Children Population - Baseline
Description: Self-reported number of Sunburns among the children of the participants in the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Sunburns
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Sunburns | 0.53 (0.02) | 0.54 (0.02) | 0.29 (0.07) | 0.20 (0.10)

72. Secondary Outcome: Sunburns - Hispanic Children Population - After Intervention
Description: Self-reported number of Sunburns among the children of the participants in the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Sunburns
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Sunburns | 0.53 (0.02) | -0.44 (0.64) | 1.21 (0.59) | -0.07 (0.11)

73. Secondary Outcome: Wearing a Hat - Hispanic Children Population - Baseline
Description: Children of participants in the Hispanic Population who wore a hat before receiving the intervention
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Participants | 1 | 1 | 2 | 7

74. Secondary Outcome: Wearing a Hat - Hispanic Children Population - After Intervention
Description: Children of participants in the Hispanic Population who wore a hat after receiving the intervention
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Participants | 0 | 0 | 2 | 4

75. Secondary Outcome: Seeking Shade - Hispanic Children Population - Baseline
Description: Self-reported number of hours of seeking shade or using an umbrella among the children of the participants in the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 0.30 (0.09) | 0.16 (0.07) | 0.32 (0.08) | 0.32 (0.07)

76. Secondary Outcome: Seeking Shade - Hispanic Children Population - After Intervention
Description: Self-reported number of hours of seeking shade or using an umbrella among the children of the participants in the Hispanic Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Hours | 0.45 (0.19) | 0.37 (0.20) | 0.52 (0.15) | 0.46 (0.13)

77. Secondary Outcome: Wearing a Shirt - Average Risk Hispanic Children Population - Baseline
Description: Children of the participants in the Hispanic Average Risk Population who reported wearing a shirt with sleeves outdoors
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27
Participants | 17 | 20

78. Secondary Outcome: Wearing a Shirt - Hispanic Children Population - After Intervention
Description: Children of the participants in the Hispanic Average Risk Population who reported wearing a shirt with sleeves outdoors, after receiving the intervention
Time Frame: 9 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27
Participants | 7 | 7

79. Secondary Outcome: Wearing a Shirt - Hispanic Children High Risk Population - Baseline
Description: Self-reported number of hours of wearing a shirt among the children of the participants in the Hispanic Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 31 | 41
Hours | 0.61 (0.09) | 0.68 (0.07)

80. Secondary Outcome: Wearing a Shirt - Hispanic Children High Risk Population - After Intervention
Description: Self-reported number of hours of wearing a shirt with sleeves outdoors among the children of the participants in the Hispanic High Risk Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 31 | 41
Hours | 0.62 (0.10) | 0.69 (0.10)

81. Secondary Outcome: Wearing Sunglasses - Hispanic Children Population - Baseline
Description: Children of the participants in the Hispanic Population who reported wearing sunglasses
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Participants | 1 | 1 | 1 | 2

82. Secondary Outcome: Wearing Sunglasses - Hispanic Children Population - After Intervention
Description: Children of the participants in the Hispanic Population who reported wearing sunglasses, after receiving the intervention
Time Frame: 9 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27 | 31 | 41
Participants | 0 | 1 | 0 | 1

83. Secondary Outcome: Wearing Sunscreen - Hispanic Children Average Risk Population - Baseline
Description: Children of the participants in the Hispanic Average Risk Population wo reported wearing sunscreen
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27
Participants | 8 | 9

84. Secondary Outcome: Wearing Sunscreen - Hispanic Children Population - After Intervention
Description: Children of the participants in the Hispanic Average Risk Population wo reported wearing sunscreen, after receiving the intervention
Time Frame: 9 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 26 | 27
Participants | 2 | 3

85. Secondary Outcome: Wearing Sunscreen - Hispanic Children High Risk Population - Baseline
Description: Self-reported number of hours of wearing sunscreen among the children of the participants in the Hispanic High Risk Population
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 31 | 41
Hours | 0.32 (0.08) | 0.39 (0.08)

86. Secondary Outcome: Wearing Sunscreen - Hispanic High Risk Children Population - After Intervention
Description: Self-reported number of hours of wearing sunscreen among the children of the participants in the Hispanic High Risk Population after receiving the intervention
Time Frame: 9 Months
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
Number analyzed (Participants) | 31 | 41
Hours | 0.29 (0.12) | 0.35 (0.13)

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected
Description: Adverse Events were not collected
Arm/Group | MC1R Average Risk- Control- Non-Hispanic White Population | MC1R Average Risk - Intervention- Non-Hispanic White Population | MC1R Higher Risk- Control - Non-Hispanic White Population | MC1R Higher Risk - Intervention- Non-Hispanic White Population | MC1R Average Risk- Control- Hispanic Population | MC1R Average Risk - Intervention- Hispanic Population | MC1R Higher Risk- Control - Hispanic Population | MC1R Higher Risk - Intervention- Hispanic Population
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03509467/Prot_SAP_000.pdf